CLINICAL TRIAL: NCT00627913
Title: Retrobulbar Injection of Anesthesia Versus Injection of Healon 5 Viscoelastic Into the Anterior Chamber in the Management of Intraoperative Floppy Iris Syndrome
Brief Title: Retrobulbar Injection of Anesthesia Versus Healon 5 in the Management of Intraoperative Floppy Iris Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to insufficient subject participation
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 27170
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Intraoperative Floppy Iris Syndrome
Keywords: Floppy Iris Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Healon 5
  Interventions: Procedure: Healon 5 injection
- 2 (Experimental): Retrobulbar Anesthetic Injection
  Interventions: Procedure: Retrobulbar anesthetic injection

INTERVENTIONS:
Procedure: Healon 5 injection — Healon 5 (2.3% Sodium hyaluronate) ophthalmic viscoelastic device will be injected into the anterior chamber as needed for pupillary dilation and adequate cataract extraction with intraocular lens placement.
  Arms: 1
Procedure: Retrobulbar anesthetic injection — 3-4cc of anesthetic (1% lidocaine/0.75% bupivicaine) will be injected with a 25 gauge needle into the extraocular muscle cone prior to patient and microscope positioning. Cataract extraction with intraocular lens placement will then proceed in standard fashion.
  Arms: 2

SUMMARY:
In this study, the investigators plan to compare the incidence and complications of intraoperative floppy iris syndrome (IFIS) during cataract surgery in patients taking tamsulosin (Flomax) and treated with retrobulbar injection of anesthesia, versus injection of Healon 5 viscoelastic into the anterior chamber.

ELIGIBILITY:
Inclusion Criteria:

* All cataract patients taking tamsulosin

Exclusion Criteria:

* Patients with any history of iridocyclitis
* Presence of iris neovascularization
* History of prior iris surgery
* Presence of traumatic cataracts
* Presence of zonular dialysis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11-11 (Actual); Study Completion 2010-11-11 (Actual)

PRIMARY OUTCOMES:
Pupil diameter after hydrodissection | 2 years

SECONDARY OUTCOMES:
Pupil diameter after nuclear removal | 2 years
Pupil diameter after cortex removal | 2 years
Pupil diameter at conclusion of surgery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A Aref, M.D., Principal Investigator — The Penn State Hershey Eye Center
Locations (1):
- Penn State Hershey Eye Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Chang DF, Osher RH, Wang L, Koch DD. Prospective multicenter evaluation of cataract surgery in patients taking tamsulosin (Flomax). Ophthalmology. 2007 May;114(5):957-64. doi: 10.1016/j.ophtha.2007.01.011. PMID 17467530